CLINICAL TRIAL: NCT05967793
Title: Effect of Kinesiology Taping on Head and Trunk Control in Children With Duchenne Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egyptian Chinese University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Noha Elserty, Assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Benha University
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio tape (Experimental): Kinesio Tape will be applied on paraspinal trunk extensors muscles for 8 weeks, changed every 3 days.
  Interventions: Other: kinesio tape
- Routine physical therapy program (Active Comparator): routine physical therapy exercise
  Interventions: Other: kinesio tape

INTERVENTIONS:
Other: kinesio tape — Kinesio Tape will be applied on paraspinal trunk extensors muscles for 8 weeks, changed every 3 days.

SUMMARY:
Muscular dystrophy (MD) is a group of muscle diseases that results in increasing weakening and breakdown of skeletal muscles over time. The disorders differ in which muscles are primarily affected, the degree of weakness, how fast they worsen, and when symptoms begin. Many people will eventually become unable to walk. Some types are also associated with problems in other organs. The muscular dystrophy group contains thirty different genetic disorders that are usually classified into nine main categories or types.

The signs and symptoms consistent with muscular dystrophy are: progressive muscular wasting, poor balance, scoliosis (curvature of the spine and the back), progressive inability to walk, waddling gait, Calf deformation, Limited range of movement, respiratory difficulty, cardiomyopathy and muscle spasms This study aimed to assess the efficacy of Kinesiology Taping on head and trunk control in patients with Duchenne muscular dystrophy

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common muscular dystrophy type in childhood. Trunk control is responsible for adaptation during weight transfers, provides and maintains the upright position of the body, organizes postural and correction reactions; and stabilizes the body to perform proximal and distal limb movements, trunk rotations, and making contact between the shoulder and pelvis. In neuromuscular diseases, the trunk is usually ignored both for assessment and treatment as muscle weakness of limbs attracts more attention. Therapists usually focus on activities of lower limb and overhead including standing, walking, climbing, and raising arms to maintain independent mobility in rehabilitation sessions. However, the trunk also gradually gets weaker as the child gets older and this may be associated with movement dysfunction of upper and lower limbs. The Kinesio Taping method is used in the rehabilitation of musculoskeletal disorders, providing either an increase or a decrease in the neural excitation of the muscle, depending on the therapeutic purpose determined after the clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. being at the age of 8-12 years
2. being able to cooperate with the instructions of physiotherapist to perform the assessments and procedures.

Exclusion Criteria:

1. having severe contracture at lower extremities
2. having another neurological and/or musculoskeletal disease diagnosis in addition to DMD. c) having a history of any lower extremity injury or orthopedic/neurologic surgery within the past 6 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
H-reflex latency and amplitude for trunk extensor | through study completion, an average of 3 months
  H- reflex will be measured by an electromyogram device, four channels electrodiagnostic system with built in amplifier will be used in prone position for levator scapulae muscles and iliocostalis lumborum muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Noha Elserty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided